CLINICAL TRIAL: NCT00166439
Title: A Phase II Trial of Oxaliplatin, Cytosine Arabinoside, Dexamethasone With Rituxan (ROAD) in Patients With Relapsed CD20+ B-Cell Non-Hodgkins Lymphoma
Brief Title: Trial of Oxaliplatin, Cytosine Arabinoside, Dexamethasone With Rituxan (ROAD) in Patients With Relapsed Non-Hodgkins Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC0485; MC0485 (Other: Mayo Clinic Cancer Center); 2328-04 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Results first posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2015-10

CONDITIONS: Lymphoma
Keywords: C04.557.386
MeSH Terms: conditions — Lymphoma | interventions — Oxaliplatin; Cytarabine; Dexamethasone; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (ROAD) (Experimental): The treatment regimen included oxaliplatin with rituximab, cytarabine, and dexamethasone (ROAD); specifically, rituximab 375 mg/m^2 IV on days 1, 8,15, and 22 (cycle 1 only); dexamethasone 40 mg PO/IV days 2-5; oxaliplatin 130 mg/m^2 IV over 2 hours on day 2; cytarabine 2000 mg/m^2 IV in 250 mL of D5W over three hours x two doses on days 2-3. The second dose of cytarabine was to be given no sooner than 12 hours after the first dose and no later than 24 hours after the conclusion of the first dose. This permitted outpatient administration if desired. Patients were provided pegfilgrastim 6 mg SC on day 4. A cycle was 21 days.
  Interventions: Drug: Oxaliplatin, Cytosine Arabinoside, Dexamethasone With Rituxan (ROAD)

INTERVENTIONS:
Drug: Oxaliplatin, Cytosine Arabinoside, Dexamethasone With Rituxan (ROAD) — rituximab 375 mg/m2 IV Weekly x 4 1 cycle only
  dexamethasone 40 mg PO/IV Days 2-5 q 21 days 2 cycles
  oxaliplatin 130 mg/m2 IV Day 2 q 21 days 2 cycles
  cytosine arabinoside 2000 mg/m2 x 2 doses IV Days 2-3 q 21 days 2 cycles
  pegfilgrastim 6 mg SQ Day 4 q21 days 2 cycles

SUMMARY:
The goals of this protocol are to determine the effect of oxaliplatin, cytosine arabinoside, and dexamethasone with Rituxan (ROAD) as treatment for patients with relapsed CD20+ B-cell non-Hodgkins lymphoma (NHL).

DETAILED DESCRIPTION:
Patients with B-cell NHL that comes back after chemotherapy are typically treated with cisplatin, high-dose cytosine arabinoside and dexamethasone (DHAP) or other platinum-based treatments. Recent studies have shown a 37% response rate in patients with large cell lymphoma to immunotherapy with Rituxan. Patients <75 years old and in otherwise good health may be candidates for high dose therapy with stem cell rescue if they have disease that remains sensitive to chemotherapy. Typically, patients are administered 2 cycles of DHAP or ICE (ifosfamide, carboplatin, and etoposide) and, if the disease responds, they proceed to high-dose therapy with stem cell support. Even patients not considered transplant candidates are also often treated with DHAP or ICE or other salvage regimens. It is likely that the response rate with DHAP alone in patients eligible for transplant is <59%. Recent studies have attempted to improve on the results from DHAP or ICE by combining them with rituxan. NCCTG has just completed a phase II trial of R-DHAP. Preliminary results of the R-ICE protocol indicate a higher response rate and longer time to progression than traditional ICE.

The problem with DHAP and ICE is that they are associated with significant side effects and specifically, with DHAP the cisplatin often causes kidney problems. In fact, some patients who are considered transplant eligible before DHAP may become transplant ineligible simply by the kidney side effects. Clearly, there is a need to improve the quality of life of patients undergoing treatment and to avoid the kidney problems.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any stage (I-IV, including those with bone marrow involvement) relapsed CD20+ B-cell non-Hodgkins lymphoma, within 5 years, with aggressive histology who have not responded to, or relapsed after, initial chemotherapy and would, if treated off-study, be treated with a platinum-containing regimen.
* CD20+ diffuse large cell, mantle cell, or transformed histologies are eligible.
* Tumor biopsy to demonstrate histology < = 6 weeks prior to registration. Computed tomography (CT) or ultrasound guided needle biopsies are acceptable as long as the pathologists can confirm histology and the CD20 positivity of the tumor.
* Measurable disease (to be considered measurable the lesion must be greater than or equal to 1.5 x 1.5 cm).
* Greater than or equal to 18 years of age.
* ECOG performance status (PS) 0, 1, or 2.
* Limited to one prior chemotherapy regimen. Antibody therapy alone or immunotherapy alone will not count as a prior regimen - only chemotherapy regimens (for example - RCHOP, CVP, etc.). External beam radiation therapy does not count as a regimen.
* The following laboratory values obtained less than or equal to 14 days prior to registration:

  * Absolute neutrophil count (ANC) greater than or equal to 1500
  * Platelets (PLT) greater than or equal to 75,000
  * Total bilirubin less than or equal to 2 mg/dL
  * Creatinine less than or equal to 1.5 x upper normal limit (UNL)

Exclusion Criteria:

* Any of the following as this regimen may be harmful to a developing fetus or nursing child:

  * Pregnant women
  * Nursing women
  * Women of childbearing potential or their sexual partners who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.)
* HIV infection.
* Prior chemotherapy or biologic therapy <= 4 weeks prior to registration .
* Persistent acute toxicities due to prior chemotherapy or biologic therapy.
* Active malignancies other than NHL.
* Central nervous system (CNS) lymphoma.
* Any of the following comorbid conditions:

  * Uncontrolled diabetes mellitus
  * Uncontrolled hypertension
  * Uncontrolled peptic ulcer disease
  * Uncontrolled infection

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-03 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick B. Johnston, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (ROAD)
Started | 50
Completed | 45
Not Completed | 5
Not completed — Ineligible | 5

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (ROAD)
Number analyzed (Participants) | 45
Age, Continuous [Median (Full Range); unit: years] | 69 [23 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate After Two Cycles of ROAD
Description: The overall response rate is defined as the percentage of patients who achieve a response after two cycles of oxaliplatin with rituximab, cytarabine, and dexamethasone (ROAD). A response was considered a Complete Response (CR) or Partial Response (PR) as defined by the NCI Sponsored International Working Group (IWG). CR: Complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms if present before therapy, and normalization of those biochemical abnormalities PR: ≥ 50% decrease in SPD of the six largest dominant nodes or nodal masses.
Time Frame: Up to 42 days
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (ROAD)
Number analyzed (Participants) | 45
percentage of patients | 58 [44 to 74]

2. Secondary Outcome: Overall Survival
Description: Survival time is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 10 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (ROAD)
Number analyzed (Participants) | 45
months | 26 [7.3 to NA] — The 95% confidence interval upper limit was not reached (below the level of detection).

3. Secondary Outcome: Progression-free Survival
Description: The progression-free survival time is defined as the time from registration to progression or death due to any cause. The distribution of progression-free survival will be estimated using the method of Kaplan-Meier. Progression is defined by the NCI Sponsored IWG as a ≥ 50% increase from nadir in the sum of the products of the greatest diameters (SPD) of any previously identified abnormal node for PRs or nonresponders and/or Appearance of any new lesion during or at the end of therapy.
Time Frame: Up to 10 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (ROAD)
Number analyzed (Participants) | 45
months | 11 [6 to 104]

ADVERSE EVENTS:
Arm/Group | Treatment (ROAD)
All-Cause Mortality (participants affected / at risk) | 26/45
Serious Adverse Events (participants affected / at risk) | 3/45
Other Adverse Events (participants affected / at risk) | 43/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (ROAD) (N=45)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (ROAD) (N=45)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 (8)
Hemoglobin decreased (Blood and lymphatic system disorders) | 19 (36)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Anal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (9)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Mucositis oral (funct/sympt) (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 33 (51)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 22 (28)
Edema limbs (General disorders) | 2 (2)
Fatigue (General disorders) | 20 (30)
Fever (General disorders) | 4 (4)
Hypersensitivity (Immune system disorders) | 1 (1)
Anal infection(gr 3/4 ANC) (Infections and infestations) | 1 (1)
Infection(gr 0/1/2 ANC) (Infections and infestations) | 1 (1)
Lip infection(unknown ANC) (Infections and infestations) | 1 (1)
Pneumonia(gr 0/1/2 ANC) (Infections and infestations) | 3 (3)
Pneumonia(gr 3/4 ANC) (Infections and infestations) | 3 (3)
Pneumonia(unknown ANC) (Infections and infestations) | 1 (1)
Sepsis(gr 0/1/2 ANC) (Infections and infestations) | 2 (2)
Skin infection(gr 3/4 ANC) (Infections and infestations) | 1 (1)
Upper respiratory infectn(gr 0/1/2 ANC) (Infections and infestations) | 1 (1)
Upr aerodigstve trct infctn(gr0/1/2 ANC) (Infections and infestations) | 1 (1)
Urinary tract infection(gr 0/1/2 ANC) (Infections and infestations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 6 (6)
Leukocyte count decreased (Investigations) | 18 (31)
Lymphocyte count decreased (Investigations) | 5 (10)
Neutrophil count decreased (Investigations) | 20 (36)
Platelet count decreased (Investigations) | 31 (65)
Anorexia (Metabolism and nutrition disorders) | 9 (11)
Blood glucose increased (Metabolism and nutrition disorders) | 9 (18)
Dehydration (Metabolism and nutrition disorders) | 6 (8)
Serum albumin decreased (Metabolism and nutrition disorders) | 3 (4)
Serum calcium decreased (Metabolism and nutrition disorders) | 2 (3)
Serum magnesium decreased (Metabolism and nutrition disorders) | 16 (21)
Serum phosphate decreased (Metabolism and nutrition disorders) | 2 (2)
Serum potassium decreased (Metabolism and nutrition disorders) | 18 (23)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 25 (47)
Recurrent laryngeal nerve palsy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Syncope vasovagal (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal mucositis (clin exam) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 2 (2)
Hypotension (Vascular disorders) | 4 (4)
Thrombosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes